CLINICAL TRIAL: NCT06858293
Title: Mental Imagery of Open and Closed Chain Exercises to Improve Quadriceps Strength Post Anterior Cruciate Ligament Reconstruction: a Feasibility Study
Brief Title: Mental Imagery to Improve Quadriceps Strength Post Anterior Cruciate Ligament Reconstruction: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HR-4875
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Mental Imagery; knee; strength; physical therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental Imagery Open Chain (Experimental): Participants will receive a paper packet with instructions to imagine themselves performing seated maximal leg extension exercises. They will be instructed to imagine the feeling of the exercise for 5 seconds, rest for 5 seconds, and repeat this 50 times with a 2-minute rest period after the 25th repetition. They will also be asked to keep track of the exercises with tallies on a table within the packet and also to record on this table if they did not complete the exercises for that day. The participant is asked to perform the exercises on five consecutive days.
  Interventions: Behavioral: Mental Imagery Open Chain
- Mental Imagery Closed Chain (Experimental): Participants will receive a paper packet with instructions to imagine themselves performing maximal standing squat exercises. They will be instructed to imagine the feeling of the exercise for 5 seconds, rest for 5 seconds, and repeat this 50 times with a 2-minute rest period after the 25th repetition. They will also be asked to keep track of the exercises with tallies on a table within the packet and also to record on this table if they did not complete the exercises for that day. The participant is asked to perform the exercises on five consecutive days.
  Interventions: Behavioral: Mental Imagery Closed Chain

INTERVENTIONS:
Behavioral: Mental Imagery Open Chain — Participants will receive a paper packet with instructions to imagine themselves performing seated maximal leg extension exercises. They will be instructed to imagine the feeling of the exercise for 5 seconds, rest for 5 seconds, and repeat this 50 times with a 2-minute rest period after the 25th repetition. They will also be asked to keep track of the exercises with tallies on a table within the packet and also to record on this table if they did not complete the exercises for that day. The participant is asked to perform the exercises on five consecutive days.
  Arms: Mental Imagery Open Chain
Behavioral: Mental Imagery Closed Chain — Participants will receive a paper packet with instructions to imagine themselves performing maximal standing squat exercises. They will be instructed to imagine the feeling of the exercise for 5 seconds, rest for 5 seconds, and repeat this 50 times with a 2-minute rest period after the 25th repetition. They will also be asked to keep track of the exercises with tallies on a table within the packet and also to record on this table if they did not complete the exercises for that day. The participant is asked to perform the exercises on five consecutive days.
  Arms: Mental Imagery Closed Chain

SUMMARY:
The goal of this clinical trial is to understand if people recovering from anterior cruciate ligament reconstruction (ACLR) surgery will complete mental imagery training and if this will improve their injured leg's strength. The main questions are:

* Will people complete a five-day mental imagery exercise schedule while in physical therapy for ACLR?
* Does mental imagery exercise help raise leg strength during ACLR recovery? Researchers will also compare if different mental imagery exercises involving leg extension or squats will change leg strength.

Participants will be asked to:

* Participate in two testing sessions to make measurements of leg function
* Complete about 10 minutes of mental imagery exercises once per day for five days at home and write down whether they complete the exercises.

ELIGIBILITY:
Inclusion Criteria:

* post anterior cruciate ligament reconstruction (ACLR) surgery
* cleared to participate in physical therapy
* currently in physical therapy related to ACLR

Exclusion Criteria:

* greater than 9 months post ACLR surgery
* history of lower back of hip pain that would limit lower limb motor testing
* current neurological condition that limits muscle strength
* history of substance abuse in the last 5 years
* any uncontrolled medical condition
* inability to follow 2-step commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention | Once per day for 5 days
  At the end of the paper packet with instructions for mental imagery exercises, there will be a survey in which participants will record whether or not they have completed the exercises. They will be instructed to fill out this form each day even if they have not done the exercise. Investigators will assess how many days participants complete the exercises.

SECONDARY OUTCOMES:
Knee Extension Strength | Pre and post 5 days of mental imagery intervention
  Maximal voluntary isometric contractions (MVICs) of the knee extensors will be conducted while the participant is seated in a Biodex Dynamometer and secured with waist and trunk straps. This will involve the participant kicking as hard as they can over 2-5 seconds. Participants will be verbally encouraged to achieve maximal force, and they will be able to see a monitor with visual instruction. Participants will be provided at least 60 seconds of rest between trials, and 5 trials will be performed. If the fifth trial produces a force more than 5% greater than any other trial, additional trials may be performed.

OTHER OUTCOMES:
Walking speed | Pre and post 5 days of mental imagery intervention
  Participants will be asked to complete the Ten Meter Walk Test which assesses self-selected and fast walking speed over the middle 6 meters of a 10-meter distance. They will walk at their self-selected and fast walking speed 3 times each over the 10-meter distance, and average speeds will be calculated.
Knee range of motion | Pre and post 5 days of mental imagery intervention
  Active and passive range of motion for knee extension and flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The investigators in this study plan to publish future findings in scientific journals and/or presentations.